CLINICAL TRIAL: NCT05606354
Title: Effects of Kinesio Taping Versus Conventional Physiotherapy in Women With Knee Osteoarthritis- A Single-Center RCT
Brief Title: Taping Versus Conventional Physiotherapy in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Aqsa Bhutto, Principal investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2644
Record Dates: First submitted 2022-10-24; First posted 2022-11-04 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis; Kinesio Taping; exercises; overweight; Female patients; degenerative disease
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity; Overweight

STUDY DESIGN:
Intervention Model Description: There are two groups: interventional and Control. Both groups will receive one standard treatment which is exercises. interventional group will receive kinesio tape and control group will not receive any kinesio tape.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Group A) (Experimental): STRECHING EXERCISES:
  A. HAMSTRING MUSCLE STRECHING.
  B. CALF MUSCLE STRECHING:
  2. STRENGTHENING EXCERCISES: 2 exercises will be performed on targeted muscle group Quadriceps. A. QUADRICEP MUSCLE (with ankle weight). B. QUADRICEP MUSCLE (straight leg raise).
  3. KNEE RANGE OF MOTION EXERCISES: (FLEXION AND EXTENSION)
  4. FUNCTIONAL EXERCISES:
  A. SIT TO STAND:
  B. CLIMBING STAIRS:
  KINESIO TAPING The following KT application techniques will be used for intervention group after identifying the goal. Goal - A: Proprioception Stimulation and Mechanical Correction Tape Technique-A: (Strip Cutting Shape: One Y-shaped + two I-shaped strips).
  Goal B: Lymphatic Correction and Muscle Correction Tape Technique-B: (Strip Cutting Shape: Two Y-shaped + two I-shaped strips).
  Interventions: Other: Intervention group
- control group (Group.B) (Other): GROUP.B - (CONTROL) - EXERCISES ONLY WITHOUT KINESIO TAPE The exercise types and dosage will be exactly the same for control group (as in experimental group (as mentioned above) But no kinesio tape will be given to this group.
  Interventions: Other: Intervention group

INTERVENTIONS:
Other: Intervention group — Experimental

SUMMARY:
The purpose of this study is to determine the effects of kinesio taping versus conventional physiotherapy in women with knee osteoarthritis.

DETAILED DESCRIPTION:
* This study will be a Randomized control trial. The calculated sample size for this study was 68 (34 in each group). To compensate the expected dropouts the sample size was increased by 15 %. Hence the final sample size will be 80 (40 in each group).
* The participants of this study will be female patients having Grade.2 knee osteoarthritis aged in between 50 to 60 years having BODY MASS INDEX (BMI) range 25-29.9(Overweight), who are being referred to Dow Ojha Physiotherapy OUT PATIENT DEPARTMENT. The subjects will be divided into 2 equal groups through Randomization Technique (Coin toss).
* Intervention group will receive regular physiotherapy exercises with Kinesio tape application, Whereas Control group will be given the same exercises without Kinesio taping.
* First assessment will be done at the baseline and second(final) will be conducted at the end of 3rd week (after 9 sessions).
* Data will be analyzed through SPSS (Statistical Package for the Social Sciences) Version-26. For mean comparison of dependent variables among Experimental and Control group Repeated Measure two-way Analysis of covariance will be performed. P-value less than 0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with knee Osteoarthritis who are being referred to Physiotherapy OPD of Dow University Ojha Campus.
* Having grade-2 Osteoarthritis (mild).)
* Aged between 50 to 60 years.
* BMI (25-29.9) -Category Overweight .
* In case of bilateral knee pain, the most painful side will be identified for intervention to see the outcome.

Exclusion Criteria:

* Total knee replacement done or any other knee surgeries.
* Rheumatoid arthritis.
* Intra articular injections received within a month.
* Knee OA -grade1(doubtful), grade3 (moderate)and grade 4 (severe).
* Altered skin sensation around the knee area.
* Having known sensitivity to tape materials.
* Underlying skin disorders.
* Recent knee trauma or fracture.

Ages: 50 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — FEMALE PATIENTS
Enrollment: 80 (Actual)
Dates: Start 2022-10-07 (Actual); Primary Completion 2024-03-10 (Actual); Study Completion 2024-03-10 (Actual)

PRIMARY OUTCOMES:
VISUAL ANALOGUE SCALE | 3 WEEKS
  USED FOR PAIN - (0CM to 10CM) 0=no pain, 10=worst pain.
THE WESTERN ONTARIO AND MCMASTER UNIVERSITIES OSTEOARTHRITIS INDEX | 3 WEEKS
  USED FOR PAIN ,STIFFNESS AND PHYSICAL FUNCTION (SCORE 0-96) 0=GOOD OUTCOME, 96=WORSE OUTCOME

CONTACTS AND LOCATIONS:
Overall Officials: aqsa bhutto, DPT, Principal Investigator — Dow University of Health Sciences
Locations (1):
- Dow institute of physical medicine and rehabilitation, Karachi, Sindh, Pakistan

REFERENCES:
- [Background] Upadhaya S, Ram CS, Kumar M, Katiyar N. EFFECT OF KINESIO TAPING AND CONVENTIONAL PHYSIOTHERAPY ON DISABILITY AND PAIN IN KNEE OSTEOARTHRITIS. Turkish Journal of Physiotherapy and Rehabilitation.;32:2.